CLINICAL TRIAL: NCT00464802
Title: A Double-Blind, Placebo-Controlled, Multiple-Dose, 2-Period Crossover Study to Evaluate the Safety and Tolerability of a New Intravenous Formulation of MOA-728 in Comparison With the Current Formulation in Healthy Subjects
Brief Title: Study Evaluating the Safety and Tolerability of a New Intravenous Formulation of MOA-728 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3200L2-1107
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: healthy; safety

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
The primary objective is to determine the safety and tolerability of the new IV formulation versus the current formulation of MOA-728 focusing on the theoretical potential for infusion-related and formulation-related complications.

ELIGIBILITY:
* A signed and dated informed consent form.
* Men or nonlactating and nonpregnant women, aged 18 to 80 years, inclusive.
* Women of nonchildbearing potential (WONCBP) must be surgically sterile (hysterectomy, oophorectomy, and/or tubal ligation) or postmenopausal for ³1 year.
* Women of childbearing potential (WOCBP) must be using an acceptable nonhormonal method of contraception (intrauterine device [IUD], diaphragm, or condom with spermicidal jelly or foam, abstinence) for a period of at least 1 month before and after dose administration.
* All women must have a negative pregnancy test result within 48 hours before the start of the first test article administration.
* Body mass index in the range of 18 to 32 kg/m² and body weight ≥50 kg.
* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).
* Subjects aged 65 to 80 years should be healthy, but may be enrolled with a chronic illness, if such illness is well controlled and does not interfere with the primary objective of the study. Certain concomitant medications will be allowed for the treatment of these conditions and are listed in the Concomitant Treatment section.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking from 48 hours before and throughout the inpatient stay.
* Have a high probability for compliance with and completion the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
IV site tolerability and urinary zinc excretion

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Phoenix, Arizona, United States